CLINICAL TRIAL: NCT06197347
Title: Web-based Nursing Intervention to Promote Physical Activity Among Older Adults With Coronary Heart Disease: Protocol for a Mixed Method Pilot Study
Brief Title: Web-based Nursing Intervention to Promote Physical Activity Among Older Adults With Coronary Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-11810
Record Dates: First submitted 2023-09-29; First posted 2024-01-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Older Adults; Web-based Intervention; Nursing; Healthy Lifestyle Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based nursing intervention (Experimental): Web-based intervention (8 sessions weekly) which includes the support of a nurse that aims to increase physical activity and quality of life for older people living with heart disease, as well as enhancing knowledge, motivation and self-efficacy.
  Interventions: Behavioral: Web-based nursing intervention : Ch@ngeons Ensemble

INTERVENTIONS:
Behavioral: Web-based nursing intervention : Ch@ngeons Ensemble — The web-based nursing intervention, named "Ch@ngeons Ensemble," was designed to increase physical activity and quality of life among older adults living with CHD. The intervention will be multicomponent, including educational content, videos, forums, goal planning, an electronic physical activity journal, and virtual written interactions with a nurse. An initial in-person meeting with the nurse will be provided to foster the older adult's commitment to the intervention and help build a relationship of trust. Throughout the intervention, the nurse will asynchronously provide counseling, feedback, and encouragement, and attempt to promote quality of life, knowledge, motivation, and self-efficacy among the older adults.

SUMMARY:
The purpose of this study is to develop and evaluate a web-based nursing intervention aimed at increasing physical activity in people aged 65 years and older with coronary heart disease.

This study aims to answer the following questions:

1. What are the needs of older adults living with coronary heart disease in terms of a web-based nursing intervention to help them increase their level of physical activity?
2. What is the acceptability (content, structure, usefulness) and feasibility (recruitment, retention, adherence, fidelity) of a web-based nursing intervention to support older adults living with coronary heart disease as they increase their level of physical activity?
3. What are the preliminary effects of the web-based nursing intervention on the physical activity level and quality of life of older adults living with coronary heart disease?
4. What are the qualitative impacts of the web-based nursing intervention as perceived by older adults on their physical activity level, quality of life, motivation, knowledge and self-efficacy?
5. How can the preliminary effects of a web-based nursing intervention, developed in response to the needs of older adults living with coronary heart disease, be illustrated by its impacts as perceived by older adults post-intervention?

A web-based nursing intervention was developed based on the needs of seniors living with coronary heart disease. 30 older adults living with heart disease will take part in the 8-week intervention. The effects of the intervention will be evaluated on the physical activity level, quality of life, knowledge, motivation and self-efficacy of older adults.

DETAILED DESCRIPTION:
Introduction: Given the high prevalence of coronary heart disease among older adults and the aging of populations, there is a need for secondary prevention interventions to help older adults become more physically active. Web-based interventions could be considered for this purpose, knowing that Internet use is growing rapidly among older adults. In addition, since older adults would appreciate developing a trusting relationship with a healthcare professional, such as a nurse, web-based interventions should include this support, which is not widely observed in the literature.

The purpose of this study is to develop and evaluate a web-based nursing intervention aimed at increasing physical activity in people aged 65 years and older with coronary heart disease.

This study aims to answer the following questions:

1. What are the needs of older adults living with coronary heart disease in terms of a web-based nursing intervention to help them increase their level of physical activity?
2. What is the acceptability (content, structure, usefulness) and feasibility (recruitment, retention, adherence, fidelity) of a web-based nursing intervention to support older adults living with coronary heart disease as they increase their level of physical activity?
3. What are the preliminary effects of the web-based nursing intervention on the physical activity level and quality of life of older adults living with coronary heart disease?
4. What are the qualitative impacts of the web-based nursing intervention as perceived by older adults on their physical activity level, quality of life, motivation, knowledge and self-efficacy?
5. How can the preliminary effects of a web-based nursing intervention, developed in response to the needs of older adults living with coronary heart disease, be illustrated by its impacts as perceived by older adults post-intervention?

Method: This study will be conducted in two phases. Phase 1 will focus on developing the intervention according to the Intervention Mapping framework, in collaboration with a team of healthcare professionals and based on the needs of older adults. In Phase 2, we will evaluate the intervention through a pilot study with a sequential explanatory design. First, a single group pre-post test will be used to assess the intervention's preliminary effects on physical activity (electronic questionnaire), quality of life (SF-36 questionnaire), knowledge (quiz), motivation and self-efficacy (visual analog scale) of 30 older adults living with coronary heart disease, as well as the feasibility of the intervention. Second, a descriptive qualitative design will employ semi-structured interviews to assess the impacts of the intervention as perceived by 8 to 12 older adults who participated in the intervention, as well as its acceptability. Non-parametric statistics and a thematic analysis will be produced. Lastly, a joint display will be used to integrate mixed data.

Discussion: The results of this study will provide insight into the development and preliminary evaluation of a web-based nursing intervention to support older adults living with coronary heart disease as they increase their physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* agreement to participate in the study about 3 months post-hospitalization for a coronary bypass graft surgery or a percutaneous coronary intervention (as motivation to change behavior would be highest during this period)
* no concurrent involvement in an intervention designed to increase their level of physical activity (e.g., a cardiac rehabilitation program, consultation with physical activity expert) during their participation in the project
* an interest in increasing their level of physical activity post-hospitalization
* fluency in French, spoken and written
* living in the greater Montreal area
* access to a computer connected to the Internet
* no cognitive impairments according to the patient record (i.e., decreased or impaired complex attention, executive functions, learning abilities, memory or social skills)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity level by the self-reported questionnaire "Electronic diary of physical activity". | Pre-intervention and immediately after the intervention.
  Self-reported questionnaire that measures the amount of physical activity performed each week in minutes.

SECONDARY OUTCOMES:
Motivation level by the digital analog scale "Motivation scale" from 1 to 10. | Pre-intervention and immediately after the intervention.
  Digital analog scale from 1 to 10 to measure motivation levels. 1 = low motivation level, 10 = high motivation level.
Self-efficacy level by the digital analog scale "Self-efficacy level" from 1 to 10. | Pre-intervention and immediately after the intervention.
  Digital analog scale from 1 to 10 to measure self-efficacy levels 1 = low self-efficacy level, 10 = high self-efficacy level.
Level of knowledge by a 5-questions multiple-choice quiz that measures knowledge of physical activity and coronary heart disease | Pre-intervention and immediately after the intervention.
  Quiz on physical activity and coronary heart disease. High score = high level of knowledge.
Quality of life level by the SF-36 questionnaire | Pre-intervention and immediately after the intervention.
  SF-36 questionnaire. High score = a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Dubé, PhD, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Univerité de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lavoie A, Dube V. Web-Based Nursing Intervention to Promote Physical Activity Among Older Adults After Coronary Revascularization: Protocol for Mixed Method Pilot Study. JMIR Res Protoc. 2025 May 21;14:e67678. doi: 10.2196/67678. PMID 40397502